CLINICAL TRIAL: NCT04611113
Title: Efficacy of Immunonutrition in Improving Tolerance to Chemoradiotherapy in Patients With Head-neck Cancer
Brief Title: Immunonutrition and Tolerance to Chemoradiotherapy in Patients With Head-neck Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Riccardo Caccialanza, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20200060578
Record Dates: First submitted 2020-10-21; First posted 2020-11-02 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer
Keywords: Immunonutrition; Chemoradiotherapy; Treatment tolerance; Nutritional counseling
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Immunonutrition Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunonutrition (Experimental): In addition to nutritional counseling, patients will receive two servings of an oral high-calorie-high-protein nutritional liquid supplement enriched in immunonutrients (Impact®). The intervention will start 10-15 days before anticancer treatment initiation and will continue until treatment termination or dropout.
  Interventions: Dietary Supplement: Immunonutrition
- Control nutritional support (Active Comparator): In addition to nutritional counseling, patients will receive two servings of an oral high-calorie-high-protein nutritional liquid supplement. The intervention will start 10-15 days before anticancer treatment initiation and will continue until treatment termination or dropout.
  Interventions: Dietary Supplement: Control Nutritional Support

INTERVENTIONS:
Dietary Supplement: Immunonutrition — In addition to nutritional counseling, patients will receive two servings of an oral high-calorie-high-protein nutritional liquid supplement enriched in immunonutrients (Impact®). The intervention will start 10-15 days before anticancer treatment initiation and will continue until treatment termination or dropout.
  Arms: Immunonutrition
Dietary Supplement: Control Nutritional Support — In addition to nutritional counseling, patients will receive two servings of an oral high-calorie-high-protein nutritional liquid supplement. The intervention will start 10-15 days before anticancer treatment initiation and will continue until treatment termination or dropout.
  Arms: Control nutritional support

SUMMARY:
The aim of the present project is to evaluate in a randomised, controlled, open-label, two parallel treatment groups pilot study, the efficacy of oral nutritional supplementation with a high-protein-high calorie mixture containing immunonutrients compared to a standard high-calorie-high-protein nutritional blend, in addition to nutritional counseling, in improving tolerance to chemoradiotherapy (CT-RT) in patients with tumours of the head and neck

DETAILED DESCRIPTION:
In a recent study, we have shown that the systematic use of oral nutritional supplements (ONS) in combination with counseling further favours the maintenance of nutrition status, the recovery of quality of life and, more importantly, improves the practicability of CT-RT. This effect would be substantially attributable to the increase in protein-energy intake associated with ONS use, but also to the possible "nutraceutical" action of omega-3 fatty acids. Therefore, modulation of the inflammatory response could play a role during cancer treatments. In this context, there is an already-known high-calorie-high-protein nutritional blend, enriched in immunonutrients (arginine, nucleotides and omega-3 fatty acids), which could also have an application in this type of patients. This mixture has proven effective in reducing the risk of post-operative complications (e.g. infections, fistulas, etc.) and the length of stay of patients undergoing major cancer surgery (abdominal and head and neck regions). Nevertheless, in oncology, there is a growing therapeutic interest in the modulation of inflammation and immunosuppression at the tumour microenvironment level.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of head-neck cancer
* indication to curative or adjuvant chemoradiotherapy
* availability to planned measurements and to written informed consent.

Exclusion Criteria:

* age <18 years
* indication to or ongoing artificial nutrition
* refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Treatment-related moderate-severe adverse events as assessed by Common Terminology Criteria for Adverse Events [CTCAE v5.0] | 9 weeks
  Difference in the incidence of grade >=3 toxicity, according to CTCAE v5.0

SECONDARY OUTCOMES:
Total chemotherapy dose | 9 weeks
  To be calculated as the percentage of chemotherapy dose administered with respect to the treatment plan
Total radiotherapy dose | 9 weeks
  To be calculated as the percentage of radiotherapy dose administered with respect to the treatment plan
Duration of treatment | 9 weeks
  To be calculated as the percentage of variation of the duration of the chemotherapy and radiotherapy compared to the planned duration
Toxicity-free survival | 9 weeks
  Difference in the time to onset of moderate-severe adverse events as assessed by CTCAE v5.0
Adherence to treatment schedule | 9 weeks
  Difference in the proportion of patients completing the treatment schedule as planned
Treatment-related adverse events as assessed by CTCAE v5.0 | 9 weeks
  Difference in the incidence of any toxicity, according to Common Terminology Criteria for Adverse Events [CTCAE v5.0]
Objective response rate | 9 weeks
  Defined as a complete response or partial response confirmed by a subsequent assessment no earlier than 2 months after the initial documentation. Response is assessed in patients with a measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST) criteria
Body weight | 9 weeks
  Change in body weight during the study
Energy intake | 9 weeks
  Change in energy intake during the study
Handgrip strength | 9 weeks
  Change in handgrip strength during the study
Skeletal muscle mass | 9 weeks
  Change in skeletal muscle mass during the study evaluated with bioimpedance vectorial analysis and computed tomography scans (C3)
Self-perceived quality of life | 9 weeks
  Change in quality of life during the study as assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire version 3.0 [EORTC QLQ-C30]
Fatigue | 9 weeks
  Change in fatigue during the study as assessed by the Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) questionnaire
Patients requiring unplanned hospitalization | 9 weeks
  The rate of patients requiring unplanned hospitalization (one or more) during the study will be calculated

OTHER OUTCOMES:
Serum levels of immunologic markers | 9 weeks
  Change in levels of soluble effectors and immuno-regulatory cells during the study

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Caccialanza, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No
Depending on a specific research question and according to a study protocol to be approved by the Ethics Committee

REFERENCES:
- [Background] Cereda E, Cappello S, Colombo S, Klersy C, Imarisio I, Turri A, Caraccia M, Borioli V, Monaco T, Benazzo M, Pedrazzoli P, Corbella F, Caccialanza R. Nutritional counseling with or without systematic use of oral nutritional supplements in head and neck cancer patients undergoing radiotherapy. Radiother Oncol. 2018 Jan;126(1):81-88. doi: 10.1016/j.radonc.2017.10.015. Epub 2017 Oct 27. PMID 29111172
- [Background] Boisselier P, Kaminsky MC, Thezenas S, Gallocher O, Lavau-Denes S, Garcia-Ramirez M, Alfonsi M, Cupissol D, de Forges H, Janiszewski C, Geoffrois L, Sire C, Senesse P; Head and Neck Oncology and Radiotherapy Group (GORTEC). A double-blind phase III trial of immunomodulating nutritional formula during adjuvant chemoradiotherapy in head and neck cancer patients: IMPATOX. Am J Clin Nutr. 2020 Dec 10;112(6):1523-1531. doi: 10.1093/ajcn/nqaa227. PMID 32936874
- [Derived] Caccialanza R, Cereda E, Klersy C, Nardi M, Masi S, Crotti S, Cappello S, Caissutti V, Brovia C, Lobascio F, Formisano E, Colombo S, Filippi AR, Bonzano E, Comoli P, Catenacci L, Alberti A, Musella V, Ferrari A, Imarisio I, Tancredi R, Monaco T, Ghi MG, Bossi P, Pedrazzoli P. The efficacy of immunonutrition in improving tolerance to chemoradiotherapy in patients with head and neck cancer, receiving nutritional counseling: study protocol of a randomized, open-label, parallel group, bicentric pilot study. Ther Adv Med Oncol. 2021 Sep 11;13:17588359211025872. doi: 10.1177/17588359211025872. eCollection 2021. PMID 34527079